CLINICAL TRIAL: NCT06119932
Title: Evaluation of One Burr Hole Evacuation for Subdural Hematoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed lotfi abdelkareem, Neurosurgical resident, Assiut University
Other Study IDs: Subdural hematoma
Record Dates: First submitted 2023-10-10; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Evacuation for subdural hematoma by one burrhole — Evacuation for subdural hematoma by one burrhole

SUMMARY:
To evaluate the outcome of one burrhole evacuation for subdural hematoma and it has the same result of traditional two burrhole

DETAILED DESCRIPTION:
* Subdural hematoma (SDH): abnormal Collection of Liquefied blood degradation underneath the dura matter (1.2.3).
* one of the most frequent types of intracranial haemorrhage, That is still associated with significant morbidity (1.4.5).
* The SDH: is a common disease in elderly Patient, and Its Incidence is highest in persons older than 70 Years of age (1.5).
* Types of Subdural hematoma(18.19)

  1- Acute: present within 48-72 hours of injury. 2. Sub-acute: manifest itself between 3-20 day. 3- Chronic (CH): produce symptoms from 3 weeks to several months after injury Risk Factors: (7.8.9.10.11.12)
  1. Trauma; mostly minor Trauma, Approximately two thirds of The Patients have suffered one. Reports exist of chronic SDH due to birth trauma in neonates.
  2. Advanced age: The elderly are at risk due to:

     1. brain atrophy, whereby The bridging veins are stretched and become more fragile.
     2. Older People tend to fall more often and Suffer minor head trauma.
     3. With increase age, The incidence of blood Thinner administration raises leading to increased risk for haemorrhage
  3. Chronic alcoholism:
  4. Gender: men, from all age groups, suffer higher rates of chsDH than woman.
  5. CoagulaPathy: Therapeutic anticoagulation and antiplatelet therapy.
  6. Medical Conditions: sepsis, hepatic failure, hemophilia, DIC and renal dialysis.
  7. Intracranial hypotension: as after ventriculoperitoneal shunt. clinical presentation (1.13)
* Symptoms of increase intra cranial pressure: Headache, Nausea, vomiting.
* Focal neurological deficit - (weakness, aphasia).
* Disturbed conscious level (DCL)
* Seizures
* Imaging investigation:

CT brain (14.15)

* Management : (1.6.16.17)

  1. Conservative: A watch, wait and re-scan Policy is usually recommended in asymptomatic or minimally symptomatic patient with a thin CHSDH.
  2. Surgical: For symptomatic (SDH) a- burr hole drainage B-twist drill drainage c- craniotomy
* prognostic factors : (2.5) 1- age of patient 2- Associated chronic diseases like hypertension, liver diseases …….Etc 3- Laboratory investigation like Hb , platlate count ,pc,and PT. 5- Hematoma thickness 6- number of burr hole : one or two burr hole

ELIGIBILITY:
Inclusion Criteria:

* Patients with subdural hematoma either unilateral or bilateral
* fit for surgery
* Chronic SDH
* Subacute SDH
* Age: patients older than 18 years old
* SEX: Both sex

Exclusion Criteria:

* Patients unfit for surgery
* Acute SDH
* subdural hyroma
* subdural empyema
* patient treated conservatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both sex Adult obove 18 years old
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
ClinicalEvaluation of evacuation for subdural hematoma by one burrhole | 72 hours post operative
  * glasgo coma scale,
  * neurological deficit,
  * clinical symptoms (seizures) .

SECONDARY OUTCOMES:
Radiological evaluation for outcome | 72 hours post operative
  Nearly gross total evacuation according to confirmation by postoperative CT brain

CONTACTS AND LOCATIONS:
Overall Officials: Shady Hassaan, Study Director — Lecturer of Neurosurgery
Locations (2):
- Egypt (2):
  - Mohammed lotfi abdelkareem, Minya, Malawi
  - Mohammed lotfi abdelkareem, Asyut